CLINICAL TRIAL: NCT02543697
Title: Adrenal Venous Sampling in Patients With Overt or Subclinical Cushings Syndrome, and Bilateral Adrenal Tumors
Acronym: AVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/2170
Record Dates: First submitted 2015-02-13; First posted 2015-09-07 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adrenal venous sampling (Experimental): Patients going trough an adrenal venous sampling to find out if hypercortisolism is uni or bilaterally produced.
  Interventions: Radiation: Adrenal venous sampling

INTERVENTIONS:
Radiation: Adrenal venous sampling — We go trough the femoral vein with a catheter up to the adrenal vein first on the left side, then on the right side. We take blood samples and analyze cortisol, metanefrin/ normetanefrin, aldosterone both from the adrenal veins and from the peripher vein. Then we use criteria from the Majo clinic to identify if the overproduction of cortisol is uni- or bilateral.

SUMMARY:
Patients with tumors in both adrenal glands and slightly elevated cortisol (subclinical Cushings syndrome) are offered to go through an adrenal venous sampling to try to quantify if the overproduction of cortisol is from one adrenal, or from both sides. If it is one-sided, the investigators offer the patient operation.

DETAILED DESCRIPTION:
Adrenal incidentalomas are quite common. About 4 % of the population have adrenal tumors that they are unknown of. Some percentage of this patients produce a little to much cortisol, but not enough to give overt Cushings syndrome. It is shown that slightly elevated cortisol production will give higher blood pressure, higher blood sugar and maybe higher BMI. For another hormone produced in the adrenal glands , aldosterone, we know that even if you have an adrenal tumor on one adrenal, you could have bilateral overproduction of the hormone.In that situations it is no need of an operation of the adrenal with the tumor. When the overproduction is unilateral it is of great value to the patient to operate the adrenal gland, and the symptoms from the hormone excess will disappear. For aldosterone Adrenal venous sampling (AVS) has been used for several years to try to determine if the hormone overproduction is one-sided or to sided. We are in this study using the same principle for cortisol overproduction.

ELIGIBILITY:
Inclusion Criteria:

* Benign tumors/adenomas in the adrenals and biochemically overproduction of cortisol

Exclusion Criteria:

* Use of steroids ( tablets, inhalations, lotions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Lateralisation of cortisol overproduction | 2 yeras
  If the ratio between cortisol in the adrenal veins is over 3,3 , it is defined as unilateral overproduction of cortisol.

SECONDARY OUTCOMES:
Biochemically and clinically normalising after treatment | 2 years
  The patients will be offered operation if the overproduction seems to be unilateral. They will then be evaluated for cortisol abnormalities , blood sugar, and hypertension i intervals of 6 months after surgery ,to see if the parameters improve. They who are not operated will be evaluated in the same way.
Verify overproduction of cortisol from the adrenals | 2 yeras
  If the ratio between cortisol in the adrenal vein and the periphery vein is over 3,3 it is defined as overproduction, and if it is over 6,5 it will probably be an adenoma.

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Ueland, MD, Principal Investigator — Haukeland Univerity Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Ueland GA, Methlie P, Jossang DE, Sagen JV, Viste K, Thordarson HB, Heie A, Grytaas M, Lovas K, Biermann M, Husebye ES. Adrenal Venous Sampling for Assessment of Autonomous Cortisol Secretion. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4553-4560. doi: 10.1210/jc.2018-01198. PMID 30137397